CLINICAL TRIAL: NCT05588206
Title: Dose-escalation by Hypofractionated Stereotactic Radiotherapy Simultaneous Integrated Boost IMRT for Brain Metastases in Non Small Cell Lung Cancer：A Phase I Study
Brief Title: Dose-escalation by Hypofractionated Stereotactic Radiotherapy for Brain Metastases in Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Hangzhou Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeHSRT
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Non Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Brain Metastases
Keywords: lung cancer; Brain Metastases; Hypofractionated Stereotactic Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Stereotactic Radiotherapy for Brain Metastases (Experimental)
  Interventions: Radiation: Hypofractionated Stereotactic Radiotherap

INTERVENTIONS:
Radiation: Hypofractionated Stereotactic Radiotherap — A standard 3+3 statistical design was employed. Three patients will initially be treated at dose level 1, 6 Gy in 5 fractions, 3 fractions a week. Dose limiting toxicities (DLT) were defined as any grade 3-5 radiation injury or any non-hematologic toxicity felt to be possibly, probably, or definitely related to radiation, identified within the evaluation period of 3 months following the completion of radiotherapy.

SUMMARY:
The objective of this trial is to assess the safety and feasibility of delivering SBRT to patients with limited BMs (less than 10 lesions of lung cancer) by establishing the maximally tolerated dose (MTD) of SABR in 5 fractions.

DETAILED DESCRIPTION:
The objective of this trial is to assess the safety and feasibility of delivering SBRT to patients with limited BMs (less than 10 lesions of lung cancer) by establishing the maximally tolerated dose (MTD) of SABR in 5 fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirmed that it was non-small cell lung cancer
* 1 to 10 brain metastases detected by magnetic resonance imaging (MRI)
* A life expectancy of >3 months according to the DS GPA.
* KPS ≥70
* Control of the primary lesions (thorax) at the time of SBRT
* 2cm<Tumor size ≤ 4 cm
* Age of 18-75 years old
* Patients must be able to undergo contrast enhanced MRI for planning
* Adequate bone marrow and organ function

Exclusion Criteria:

* other malignant tumors
* Prior surgery to brain metastasis
* Prior brain radiotherapy
* Non-small cell lung cancer with more than 10 brain metastases detected by MRI
* Contraindication to receiving radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD | 1 years
  maximum tolerated dose

SECONDARY OUTCOMES:
ARE | 2 years
  adverse radiation effect
iPFS | 2 years
  intracranial progression-free survival defines as intervals from treatment to intracranial disease progression or death
OS | 2 years
  overall survival (OS) intervals from treatment to death or last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Kaicheng Pan, Hangzhou, China